CLINICAL TRIAL: NCT02235688
Title: An Open-Label Phase 1b Study to Investigate the Preliminary Safety and Activity of Aldoxorubicin Plus Gemcitabine in Subjects With Metastatic Solid Tumors
Brief Title: Study to Investigate the Safety and Activity of Aldoxorubicin Plus Gemcitabine in Subjects With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P1-MTD-03
Record Dates: First submitted 2014-08-15; First posted 2014-09-10 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2017-06

CONDITIONS: Metastatic Solid Tumors
Keywords: aldoxorubicin; INNO-206; solid tumors; gemcitabine; phase 1
MeSH Terms: interventions — DOXO-EMCH; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aldoxorubicin (Experimental)
  Interventions: Drug: aldoxorubicin; Drug: gemcitabine

INTERVENTIONS:
Drug: aldoxorubicin — administered at 170 mg/m2 by intravenous infusion (IVI) on Day 1 every 21 days plus 900 mg/m2 gemcitabine on Days 1 and 8 every 21 days.
  Other Names: INNO-206
Drug: aldoxorubicin — administered at 250 mg/m2 by intravenous infusion (IVI) on Day 1 every 21 days plus 900 mg/m2 gemcitabine on Days 1 and 8 every 21 days.
  Other Names: INNO-206
Drug: aldoxorubicin — administered at 350 mg/m2 by intravenous infusion (IVI) on Day 1 every 21 days plus 900 mg/m2 gemcitabine on Days 1 and 8 every 21 days.
  Other Names: INNO-206
Drug: gemcitabine

SUMMARY:
This is a Phase 1 study to investigate the safety and activity of aldoxorubicin plus gemcitabine in Subjects with solid tumors.

DETAILED DESCRIPTION:
An open-label Phase 1b study to investigate the preliminary safety and activity of aldoxorubicin plus gemcitabine in subjects with metastatic solid tumors administered at doses of 170, 250 or 350 mg/m2 by intravenous infusion (IVI) on Day 1 every 21 days plus 900 mg/m2 gemcitabine on Days 1 and 8 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15-80 years, male or female.
2. Advanced, unresectable, metastatic solid tumor that has either relapsed or was refractory to treatment with at least 1 prior chemotherapy or immunotherapy regimen and for which no standard approved therapy exists.
3. Progressive disease (PD) < 6 months prior to enrollment.
4. Capable of providing informed consent and complying with trial procedures.
5. ECOG PS 0-2 (Appendix B).
6. Life expectancy >12 weeks.
7. Measurable tumor lesions according to RECIST 1.1 criteria.
8. Women must not be able to become pregnant (eg post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
9. Males and their female partner(s) of child-bearing potential must use 2 forms of effective contraception (see Inclusion 8 plus condom or vasectomy for males) from the last menstrual period of the female partner during the study treatment and for 6 months after the final dose of study treatment.
10. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
11. Geographic accessibility to the site that ensures the subject will be able to keep all study-related appointments.

Exclusion Criteria:

1. Prior exposure to >5 cycles or 375 mg/m2 of either doxorubicin or Doxil®.
2. Chemotherapy, palliative surgery and/or radiation treatment less than 30 days prior to enrollment.
3. Exposure to any investigational agent within 30 days of enrollment.
4. CNS metastases that are symptomatic.
5. History of other malignancies except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix unless documented free of cancer for ≥5 years.
6. Laboratory values: Screening serum creatinine >1.5×ULN, ALT >3×ULN, or >5×ULN if liver metastases are present, total bilirubin >3×ULN, ANC <1,500/mm3, platelet concentration <100,000/mm3, hematocrit level <25% for females or <27% for males, coagulation tests (PT, PTT, INR) >1.5×ULN, and albumin <2.0 g/dL.
7. Clinically evident CHF > class II of the NYHA guidelines (Appendix D).
8. Current serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V (Appendix F).
9. Baseline QTc >470 msec and/or previous history of QT prolongation while taking other medications. Concomitant use of medications associated with a high incidence of QT prolongation is not allowed (Appendix G).
10. History or signs of active coronary artery disease with or without angina pectoris.
11. Serious myocardial dysfunction defined scintigraphically (eg MUGA, myocardial scintigram) or ultrasound determined absolute LVEF <45% of predicted.
12. History of HIV infection.
13. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
14. Major surgery within 21 days prior to enrollment.
15. Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
16. Any condition that is unstable and could jeopardize the subject's participation in the study.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety Measures | 14 months
  The primary objective of this study is to determine the preliminary safety of administration of aldoxorubicin in combination with gemcitabine in subjects with metastatic solid tumors as measured by the frequency and severity of adverse events (AEs), abnormal findings on physical examination, laboratory tests, vital signs, echocardiograms (ECHO) or multiple-gated acquisition (MUGA) scans, electrocardiogram (ECG) results, and weight.

SECONDARY OUTCOMES:
Tumor Response | 17 months
  The secondary objective of this study is to evaluate the activity of aldoxorubicin in combination with gemcitabine in this population, assessed by overall response rate (ORR) and progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, M.D., Study Director — CytRx Coporation
Locations (2):
- United States (2):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - Sarcoma Oncology Center, Santa Monica, California